CLINICAL TRIAL: NCT05805878
Title: Knowledge, Attitudes and Practices Regarding Tuberculosis Among Physicians in Assiut City
Brief Title: KAP Regarding Tuberculosis Among Physicians in Assiut City
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Abd Elkareem Mariae Mohamed, Demonstrator, Assiut University
Other Study IDs: KAP regarding Tuberculosis
Record Dates: First submitted 2023-03-22; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To Strengthen tuberculosis education and awareness among physicians in Assiut city in the framework of national tuberculosis control program.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains a major global health problem. According to the World Health Organization (WHO), an estimated global total of 10.6 million people fell ill with TB in 2021, equivalent to 134 cases per 100 000 populations. About 1.5 million people die from TB each year - making it the 13th leading cause of death worldwide . Until the coronavirus (COVID-19) pandemic, TB was the leading cause of death from a single infectious agent, ranking above human immunodeficiency virus (HIV). TB is present in all countries but it is highly prevalent among the low socioeconomic section of the population and marginalized sections of the community .

TB is an infectious bacterial disease caused by Mycobacterium tuberculosis (Mtb), which is transmitted between humans through the respiratory route and most commonly affects the lungs, but can damage any tissue . Only about 10 percent of individuals infected with Mtb progress to active TB disease within their lifetime; the remainder of persons infected successfully contain their infection. One of the challenges of TB is that the pathogen persists in many infected individuals in a latent state for many years and can be reactivated to cause disease. According to WHO, approximately one-quarter of the world's population is latently infected with Mtb . The risk of progression to TB disease after infection is highest soon after the initial infection and increases dramatically for persons co-infected with HIV or other immune-compromising conditions .

TB is a curable and preventable disease. TB drugs are administered in different combinations of four first-line drugs which form the core of treatment regimens in the initial treatment phase of 6-9 months. Several reasons account for the failure of TB therapy such as (i) late diagnosis, (ii) lack of timely and proper administration of effective drugs, (iii) long treatment duration, (iv) non adherence to drug regimen and (v) evolution of drug-resistant TB strains. Drug-resistant TB(DR-TB) poses a significant challenge to TB therapy and control programs .

In 2014 and 2015, all Member States of WHO and the United Nations (UN) committed to ending the TB epidemic, through their adoption of WHO's End TB Strategy and the UN Sustainable Development Goals (SDGs). The UN SDGs include ending the TB epidemic by 2030 under Goal 3. WHO's End TB Strategy aims to reduce TB deaths by 90% and cut new cases by 80% between 2015 and 2030, and ensure that no family is burdened with catastrophic health expenditure due to TB.

In Egypt TB is still a health problem, which affects the young active age group with pulmonary TB more in Lower Egypt, whereas extrapulmonary cases were more in Upper Egypt, especially in the rural community . Egypt is ranked among the mid-level incidence countries and according to a WHO estimation of the TB burden in 2019, the incidence of TB was 12 per 100 000 inhabitants . The Ministry of Health and Population (MOHP) has established the National Tuberculosis Control Program(NTP) in 1979 .

The COVID-19 pandemic has undone decades of progress in the fight against TB. Globally, the estimated number of deaths from TB increased between 2019 and 2021, reversing years of decline between 2005 and 2019. The burden of DR-TB is also estimated to have increased between 2020 and 2021, with 450 000 new cases of rifampicin-resistant TB . The most obvious and immediate impact was a large global drop in the reported number of people newly diagnosed with TB. Reductions in the reported number of people diagnosed with TB in 2020 and 2021 suggest that the number of people with undiagnosed and untreated TB has grown, resulting in an increased number of TB deaths and more community transmission of infection and increased numbers of people developing TB .

Healthcare workers (HCWs) play a fundamental role in the global fight against TB . Adequate basic knowledge about TB enables the physician to suspect and deal with a TB case, whereas insufficient knowledge will lead to either escaping suspicion or improper dealing with a TB case. The delayed proper diagnosis and management of TB will cause spreading of TB and facilitate the development of resistance to anti-TB drugs .

Worldwide, many studies found that HCWs have important knowledge gaps in relation to TB diagnosis, treatment and infection prevention and control; have some negative attitudes and stigma connected with the disease; and engage in poor practices, all of which contribute to their increased risk of infection and negative impacts on patients and the community .

In Egypt, previous studies illustrated lower basic knowledge of the studied primary health care (PHC) physicians about TB. In Gharbia Governorate , the mean of satisfactory basic knowledge was 49.6%. Similar results were detected in Menofya Governorate and in Qalyubia Governorate, where the means of satisfactory basic knowledge of the studied physicians about TB were 54.5% and 48.2% respectively. Other study in Behaira Governorate reported a mean of 63% for physicians' knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Non specialist Physicians working and providing medical care in primary health care units and Hospitals in Assiut city.

Exclusion Criteria:

* specialist Physicians

Ages: 26 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: Non specialist Physicians working and providing medical care in primary health care units and Hospitals in Assiut city.
Sampling Method: Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
To assess knowledge, attitudes and practices (KAP) on tuberculosis among physicians working in Assiut city. | 3 years
  questionnaire will be used to assess this outcome measure.

SECONDARY OUTCOMES:
To explore the factors associated with the physicians' knowledge, attitudes and practices regarding tuberculosis. | 3 years
  questionnaire will be used to assess this outcome measure

REFERENCES:
- [Background] Singh R, Dwivedi SP, Gaharwar US, Meena R, Rajamani P, Prasad T. Recent updates on drug resistance in Mycobacterium tuberculosis. J Appl Microbiol. 2020 Jun;128(6):1547-1567. doi: 10.1111/jam.14478. Epub 2019 Oct 29. PMID 31595643
- [Background] Vigenschow A, Edoa JR, Adegbite BR, Agbo PA, Adegnika AA, Alabi A, Massinga-Loembe M, Grobusch MP. Knowledge, attitudes and practices regarding tuberculosis amongst healthcare workers in Moyen-Ogooue Province, Gabon. BMC Infect Dis. 2021 May 27;21(1):486. doi: 10.1186/s12879-021-06225-1. PMID 34039304